CLINICAL TRIAL: NCT05258253
Title: Effects of High Intensity Aerobics and Pelvic Clock Exercises in Primary Dysmenorrhea
Brief Title: Effects of HIA and PCE in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0505 Asmaa Qamar
Record Dates: First submitted 2022-02-20; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Primary Dysmenorrhea
Keywords: high intensity aerobics; primary dysmenorrhea; aerobics; painful menstruation
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high intensity aerobics (Experimental): "London bridges (8mins)","Jumping lunges(8mins)","Mountain climbers(8mins)","Quadruped bent knee hip extension (8mins)"
  Interventions: Other: High intensity aerobics
- pelvic clock exercises (Active Comparator): Lie with your back on the floor in a neutral position with your legs bent and toes facing forward. Subject begin with gentle movements from 12 to 6 o'clock, as instructed to move from 3 o'clock to 9 o'clock. Then move in a clockwise manner from 12 to 3 to 6 to 9 and then back to 12 o' clock.
  Interventions: Other: Pelvic clock exercises

INTERVENTIONS:
Other: High intensity aerobics — "London bridges (8mins)" "Jumping lunges(8mins)" "Mountain climbers(8mins)" "Quadruped bent knee hip extension (8mins)"
  Arms: high intensity aerobics
Other: Pelvic clock exercises — Lie with your back on the floor in a neutral position with your legs bent and toes facing forward. Subject begin with gentle movements from 12 to 6 o'clock, as instructed to move from 3 o'clock to 9 o'clock. Then move in a clockwise manner from 12 to 3 to 6 to 9 and then back to 12 o' clock.
  Arms: pelvic clock exercises

SUMMARY:
The main purpose of study is to manage the unpleasant pain suffered by females during Mensturation. The aim of this study is to guide physiotherapist that how to apply these exercises to manage dysmenorrhea.

DETAILED DESCRIPTION:
There are less research on effectiveness of pelvic clock exercises in dysmenorrhea they are very less evidence and less documented in literature.. Although there are many researches on high intensity aerobics.Previous researches only have lierature about aerobics.So to address this literature gap, conduct a prospective randomized controlled trial to investigate the effects of high intensity aerobics and pelvic clock exercises in primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Girls aged 17-23 years with regular menstrual cycle
* Unmarried girls

Exclusion Criteria:

* Athletes, Married women,
* Girls who were regularly exercising
* Having any pelvic pathology, abnormal menstrual cycle.

Ages: 17 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — only females
Enrollment: 28 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-11-13 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | last 1 day
  Scores are recorded by making a mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

SECONDARY OUTCOMES:
DASS 21 | last 1 day
  DASS-21 scale contains 7 items, divided into subscales with similar content.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Aabroo, PPDPT, Principal Investigator — Riphah International University
Locations (1):
- Rasheeda gynae hospital, Hafizabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No